CLINICAL TRIAL: NCT01709123
Title: Ketosis, Vascular Inflammation, and Its Therapy (Chromium Supplementation) in Diabetic Patients
Brief Title: Effects of Micronutrient (Chromium) Supplementation on Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-08-028; 3R01DK072433-03S1 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Juvenile Onset; Cardiovascular Diseases; Hyperglycemia; Hyperketonemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Hyperglycemia; Ketosis | interventions — chromium nicotinic acid complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo supplementation in pill form for 3 months following randomization after a placebo run-in period.
  Interventions: Drug: placebo
- chromium niacinate (Experimental): Chromium niacinate supplementation (200ug or 500ug/day) in pill form for 3 months following randomization after a placebo run-in period
  Interventions: Drug: chromium niacinate

INTERVENTIONS:
Drug: chromium niacinate — 200ug or 500ug supplementation in pill form
  Arms: chromium niacinate
Drug: placebo — Placebo pill for chromium niacinate
  Arms: placebo

SUMMARY:
6-8% of USA population has diabetes. Intensive blood glucose control dramatically reduces the devastating complications that result from poorly controlled diabetes. However, for many patients, achievement of tight glucose control is difficult with current regimens. Trivalent chromium, the form found in foods and dietary supplements, is believed to be safe. Our preliminary studies have reported that chromium supplementation inhibits the increase in pro-inflammatory cytokines (tumor necrosis factor-alpha and interleukin-6; TNF-alpha and IL-6) secretion levels caused by high glucose levels in cultured monocytic cells. Similarly, animal studies have shown that chromium niacinate supplementation lowered blood levels of glycemia and pro-inflammatory cytokines in streptozotocin-treated diabetic rats. Cytokines are proteins that are secreted by monocytes and other cells in response to various stimuli, such as infection. Some of the cytokines are known to regulate insulin sensitivity and elevated level of these cytokines in blood may accelerate clogging of arteries. Thus, chromium supplementation may increase insulin sensitivity and glycemic control in diabetic patients, and may prevent the development of cardiovascular disease in diabetic patients. Given the enormous public health cost of diabetes, the prospect of being able to use a relatively low-cost dietary supplement, such as chromium, as an adjuvant therapy to help in achieving normal blood glucose level merits further study.

We will examine the effects of placebo and chromium niacinate supplementation on the fasting glucose, cholesterol, triglycerides, and markers of vascular disease in blood of diabetic patients. We will determine these above parameters at baseline and after the 1, 2 and 3 months of supplementation in diabetic patients. The long-term objective is to explore the efficacy of chromium as an adjuvant treatment for better glycemic control, prevent the development of cardiovascular disease (CVD), and improve the life expectancy in diabetic population.

Chromium supplements are widely used by the public and are available in many stores, such as Wal-mart, Walgreens, and many other food and drug stores. Chromium is an essential trace metal and micronutrient present in wide variety of vegetables. Niacin is a vitamin B6, an essential vitamin for our body. This study plans to use chromium niacinate, a complex of chromium and niacin. Chromium niacinate is considered a nutrient.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes mellitus
* Participants between the ages of 8 and 21

Exclusion Criteria:

* Subjects with sickle cell disease, renal or liver disease
* Serum positive pregnancy test or breastfeeding
* Participants unwilling/unable to take supplements in pill form
* Participants taking prescription medication or supplements

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2007-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sushil K Jain, Ph.D., Principal Investigator — Louisiana State University Health Sciences Center in Shreveport
Locations (1):
- Louisiana State University Health Sciences Center in Shreveport, Shreveport, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Chromium Niacinate
Started | 31 | 31
Completed | 22 | 22
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Population: The original number of enrolled participants was 62. 18 participants withdrew from the study, leaving 44 participants to remain, with 22 participants in each category.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Chromium Niacinate | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Level
Description: Measuring levels of glycemia (fasting glucose) in blood of patients in the placebo group and the chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
mg/dL
  Baseline Figures | 172.39 (20.641) | 212.85 (21.153)
  Figures:16 weeks | 164.47 (16.187) | 191.25 (21.363)

2. Primary Outcome: Blood Glucose Levels
Description: Measuring levels of glycemia (HbA1c) in blood patients in the placebo group and the chromium supplement group.
Time Frame: Assessed for 16 weeks with five measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks). 16 weeks reported.
Measure: Mean (Standard Error); unit: mmol/mol
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
mmol/mol
  Baseline Figures | 9.5667 (0.4708) | 9.7368 (0.4888)
  Figures: 16 weeks | 9.2267 (0.4396) | 9.5606 (0.4839)

3. Secondary Outcome: Lipid Levels
Description: Measuring levels of TG (triglycerides), LDL and HDL-cholesterol in blood of patients in the placebo group and the chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
mg/dL
  Baseline Cholesterol values | 165.50 (10.095) | 160.42 (7.1301)
  Cholesterol values:16 weeks | 158.87 (7.6000) | 164.78 (9.1092)
  Baseline HDL values | 50.944 (2.7871) | 53.842 (3.1122)
  HDL values:16 weeks | 49.733 (2.6806) | 54.889 (3.1425)
  Baseline LDL values | 96.000 (7.7147) | 87.579 (5.5442)
  LDL values:16 weeks | 93.867 (7.2170) | 93.556 (6.4409)
  Baseline triglyceride values | 92.333 (10.538) | 91.105 (13.914)
  Triglyceride values:16 weeks | 77.200 (6.0688) | 81.722 (14.557)

4. Secondary Outcome: Blood Levels of Cytokines/Inflammatory Biomarkers
Description: Measuring levels of reactive oxygen species (ROS) in blood of patients in the placebo group and chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: mean fluorescent unit
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
mean fluorescent unit
  Baseline ROS values | 53587.3 (1471.25) | 51877.2 (977.774)
  ROS values:16 weeks | 56864.8 (1474.31) | 53577.0 (2970.86)

5. Secondary Outcome: Blood Levels of Cytokines/Inflammatory Biomarkers
Description: Measuring levels of Interleukin-6 (IL-6) in blood of patients in the placebo group and chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
ug/mL
  Baseline Interleukin-6 Values | 1.6795 (0.1801) | 1.7754 (0.1848)
  Interleukin-6 Values: 16 weeks | 2.0290 (0.4057) | 2.0000 (0.3527)

6. Secondary Outcome: Blood Levels of Cytokines/Inflammatory Biomarkers
Description: Measuring levels of C reactive protein (CRP) in blood of patients in the placebo group and chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
ug/mL
  Baseline CRP values | 185.20 (9.8926) | 186.48 (7.6407)
  CRP values: 16 weeks | 182.98 (9.5580) | 185.11 (8.6807)

7. Secondary Outcome: Blood Levels of Cytokines/Inflammatory Biomarkers
Description: Measuring levels of Leptin in blood of patients in the placebo group and chromium supplement group.
Time Frame: Assessed for 16 weeks with 5 measurements. (0 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks), 16 weeks reported.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Placebo | Chromium Niacinate
Number analyzed (Participants) | 22 | 22
ug/mL
  Baseline Leptin values | 16.715 (4.2746) | 16.263 (3.3631)
  Leptin: 16 weeks | 15.885 (4.1824) | 14.776 (3.1102)

ADVERSE EVENTS:
Arm/Group | Placebo | Chromium Niacinate
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes